CLINICAL TRIAL: NCT06883864
Title: Efficacy and Safety of Catheter abLation in patiEnts With seVere Atrial Functional Mitral regurgiTation and pErsistent Atrial Fibrillation: a Randomized Controlled Trial (ELEVATE-AF)
Brief Title: Efficacy and Safety of Catheter abLation in patiEnts With seVere Atrial Functional Mitral regurgiTation and pErsistent Atrial Fibrillation: a Randomized Controlled Trial
Acronym: ELEVATE-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Chang sheng Ma, Director of Cardiology Department, Beijing Anzhen Hospital, Capital Medical University, Director of Beijing Cardiovascular Disease Prevention Office and Director of Department of Cardiology in Capital Medical University, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025KLS10; 2022YFC3601303 (Other Grant/Funding Number: the National Key Research and Development Program of China)
Record Dates: First submitted 2025-03-11; First posted 2025-03-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation (AF); Catheter Ablation; Atrial Functional Mitral Regurgitation
Keywords: atrial fibrillation; mitral regurgitation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation; Mitral Valve Insufficiency | interventions — Catheter Ablation; Dosage Forms; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Catheter ablation plus medication group (Experimental): All patients assigned to the catheter ablation group will receive AF catheter ablation and receive the same medical therapy as the control group.
  Interventions: Procedure: Catheter ablation plus medication; Procedure: (ELEVATE-AF X) experimental group
- Medication group (Active Comparator): All patients should receive guideline-directed medical therapy, anticoagulation, and rate control with medications according to the guidelines.
  Interventions: Drug: Medication; Procedure: (ELEVATE-AF X) control group

INTERVENTIONS:
Procedure: Catheter ablation plus medication — All patients will receive atrial fibrillation catheter ablation. They also should receive guideline-directed medical therapy, anticoagulation, and rate control with medications according to the guidelines.
  Arms: Catheter ablation plus medication group
Drug: Medication — Patients will receive guideline-directed medical therapy, anticoagulation, and rate control according to the guidelines for the management of AF and heart failure.
  Arms: Medication group
Procedure: (ELEVATE-AF X) experimental group — Subsequent ablations may be considered for patients with recurrence，and the medical therapy for ELEVATE-AF X is identical to that of the ELEVATE-AF trial.
  Arms: Catheter ablation plus medication group
Procedure: (ELEVATE-AF X) control group — All patients could receive catheter ablation if the procedure is needed, and the medical therapy for ELEVATE-AF X is identical to that of the ELEVATE-AF trial.
  Arms: Medication group

SUMMARY:
Atrial fibrillation (AF) leads to atrial functional mitral regurgitation (MR) through mechanisms including mitral annular dilatation, systolic leaflet motion distance alteration, and contractility decrease. Compared with primary MR, atrial functional MR due to AF and other diseases tends to have a worse prognosis, with a higher risk of death and heart failure hospitalization. MR and AF co-exist and exacerbate left atrial dysfunction, further causing worse cardiac dysfunction, valvular regurgitation, and aggravating prognosis.

The best therapy for secondary MR is unclear because MR is only one component of the disease, and restoration of mitral valve competence is not curative. Catheter ablation improves symptoms and cardiac function in patients with AF, reduces risks of AF recurrence and hospitalization, as well as increases quality of life. For patients with AF combined with functional moderate-to-severe MR, previous observational studies have found that the severity of MR significantly reduced after taking catheter ablation to restore sinus rhythm. We hypothesized that catheter ablation would significantly improve the severity of MR in patients with severe atrial functional MR combined with persistent AF compared with drug therapy alone.

DETAILED DESCRIPTION:
The ELEVATE-AF is a multi-center, open-label, parallel design, randomized controlled trial. Eligible subjects will be randomized in a 1:1 ratio to the catheter ablation combined with drug group or to the drug-alone group. A total of 146 patients with persistent atrial fibrillation and severe atrial functional mitral regurgitation (MR) (severity of moderate-to-severe [3+] or severe [4+]) will be enrolled at up to 17 investigational sites in China. The enrollment period is estimated to last approximately 18 months. The primary endpoint is the proportion of patients with residual MR of moderate [2+] or less assessed by transthoracic echocardiography at 3 months. MR severity is confirmed by the Echocardiography Core Lab according to the American Society of Cardiac Ultrasound criteria (mitral effective regurgitant orifice area [EROA)]≤20 mm2). The secondary endpoints evaluate: (i)all-cause mortality; (ii)cardiovascular hospitalization; (iii)undergoing interventional or surgical treatment of mitral valve; (iv)heart failure hospitalization or emergency room visit; (v)change in scores on the Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) Questionnaire, and the 5-level EQ-5D version (EQ-5D-5L); (vi) freedom from any documented atrial arrhythmias lasting more than 30 seconds and atrial fibrillation burden. The safety endpoints include: (i)perioperative surgical complications (within 30 days after catheter ablation procedure); (ii)major bleeding (ISTH definition); (iii)stroke and systemic embolism.

As an extension of the ELEVATE-AF trial, ELEVATE-AF X study will conducted after 3-month follow-up of ELEVATE-AF. The ELEVATE-AF X study is designed as a prospective, multi-center, continued access registry study. The objective of the this study is to validate the long-term outcomes of catheter ablation procedure in patients with persistent AF and severe atrial functional MR. All patients will receive catheter ablation if the procedure is needed, and the medical therapy for ELEVATE-AF X is identical to that of ELEVATE-AF trial. Active follow-up of patients will be performed through 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were required to have moderate-to-severe or greater (≥3+) atrial functional mitral regurgitation assessed by transthoracic echocardiography within 14 days before randomization. Mitral regurgitation severity was graded by an echocardiography core-lab based on the American Society of Echocardiography criteria, specifically an effective regurgitant orifice area (EROA) ≥30 mm²
2. Age 18-80 years
3. Persistent atrial fibrillation diagnosed by electrocardiogram
4. Left ventricular ejection fraction ≥50% assessed by transthoracic echocardiography within 14 days before randomization(confirmed by the echocardiography core-lab)
5. Left ventricular end-diastolic internal diameter ≤60 mm and left atrial anterior- posterior diameter ≤60 mm in echocardiographic parasternal long-axis view within 14 days before randomization(confirmed by the echocardiography core-lab)
6. Within 14 days before randomization, patients must be treated to ensure the absence of fluid retention and to maintain an average heart rate below 110 bpm.
7. Agree to undergo catheter ablation and be able to undergo follow-up as required.

For the ELEVATE-AF X study: Subjects have to meet the ELEVATE-AF study eligibility criteria to be registered in the ELEVATE-AF X study.

Exclusion Criteria:

1. paroxysmal atrial fibrillation, atrial fibrillation secondary to an apparently reversible cause, or with history of previous ablation;
2. primary mitral valve pathology, including calcification, sclerosis, prolapse, flail, tendon cable rupture, valve degeneration, infective endocarditis, rheumatic lesions, or ischemic lesions;
3. history of previous mitral valve surgery or transcatheter manipulation;
4. mitral valve orifice area <4 cm2;
5. aortic valve disease requiring surgical or transcatheter intervention;
6. untreated clinically significant coronary artery disease requiring revascularization;
7. history of previous myocardial infarction;
8. previous definitive diagnosis of cardiomyopathies such as dilated cardiomyopathy, hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, arrhythmogenic cardiomyopathy, and infiltrative cardiomyopathies (e.g., amyloidosis, hemochromatosis, and nodular disease)
9. echocardiographic evidence of intracardiac mass or thrombus;
10. implant of cardiac device (pacemaker, implantable cardioverter defibrillator, cardiac resynchronization therapy device, or left atria appendage closure);
11. hemodynamic instability requiring cardiac assist devices, intra-aortic balloon pump (IABP), or other hemodynamic support;
12. any percutaneous cardiac intervention (percutaneous coronary intervention, transcatheter aortic valve replacement, etc.) within the 30 days prior to randomization,
13. any cardiac surgery within the 6 months prior to randomization;
14. active infections requiring current antibiotic therapy;
15. a known hypersensitivity or contradiction to procedure medications which cannot be adequately managed medically;
16. contraindication to appropriate anti-coagulation therapy;
17. chronic obstructive pulmonary disease (COPD) requiring continuous home oxygen therapy or chronic oral steroid therapy;
18. acute cerebrovascular accident within 30 days prior to randomization or Modified Rankin Score ≥ 4;
19. symptomatic severe carotid stenosis (>70% by ultrasound);
20. other planned surgical or interventional procedures within the next 3 months;
21. liver failure;
22. renal failure or dialysis status;
23. pregnant or planning pregnancy within the next 3 months;
24. life expectancy < 12 months (e.g., advanced malignant tumors);
25. currently participating in other interventional studies;
26. circumstances that, in the judgment of the researcher, make participation in this study unsuitable.

For the ELEVATE-AF X study: Subjects who have any contraindications to ELEVATE-AF study and are not capable of performing ELEVATE-AF study per investigator's assessment should not be registered in the ELEVATE-AF X study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of patients with residual MR of moderate [2+] or less assessed by transthoracic echocardiography at 3 months. | 3 month
  The primary endpoint is the proportion of patients with residual MR of moderate [2+] or less assessed by transthoracic echocardiography at 3 months. MR severity is confirmed by the Echocardiography Core Lab according to the American Society of Cardiac Ultrasound criteria (mitral effective regurgitant orifice area [EROA)]≤20 mm2).

SECONDARY OUTCOMES:
all-cause mortality | 3 month
cardiovascular hospitalization | 3 month
undergoing interventional or surgical treatment of mitral valve | 3 month
heart failure hospitalization or emergency room visit | 3 month
Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) score change between baseline and 3 month | 3 month
  Quality of life assessed by AFEQT questionaire
EuroQoL 5-Dimension 5-Level (EQ-5D-5L) score change between baseline and 3 month | 3 month
  Quality of life assessed by EQ-5D-5L scale
freedom from any documented atrial arrhythmias lasting more than 30 seconds and atrial fibrillation burden | 3 month
(ELEVATE-AF X) the proportion of patients with residual MR of moderate [2+] or less assessed by transthoracic echocardiography | 12 month
(ELEVATE-AF X) all-cause mortality | 12 month
(ELEVATE-AF X) cardiovascular hospitalization | 12 month
(ELEVATE-AF X) undergoing interventional or surgical treatment of mitral valve | 12 month
(ELEVATE-AF X) heart failure hospitalization or emergency room visit | 12 month
(ELEVATE-AF X) Atrial Fibrillation Effect on QualiTy-of-life (AFEQT) score change between baseline and 12 month | 12 month
  Quality of life assessed by AFEQT questionaire
(ELEVATE-AF X) EuroQoL 5-Dimension 5-Level (EQ-5D-5L) score change between baseline and 12 month | 12 month
  Quality of life assessed by EQ-5D-5L scale
(ELEVATE-AF X) freedom from any documented atrial arrhythmias lasting more than 30 seconds and atrial fibrillation burden | 12 month

OTHER OUTCOMES:
perioperative procedural complications | 3 months
major bleeding (ISTH definition) | 3 months
stroke and systemic embolism | 3 months
(ELEVATE-AF X) major bleeding (ISTH definition) | 12 month
(ELEVATE-AF X) stroke and systemic embolism | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, MD, Principal Investigator — Beijing Anzhen Hospital; Caihua Sang, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No